CLINICAL TRIAL: NCT05278949
Title: A Novel Technique of Re-fixating Dislocated Scleral Fixing Intra-ocular Lens
Brief Title: Re-fixating Dislocated Scleral Fixing Intra-ocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omer Othman Abdullah (Other)
Responsible Party: Sponsor-Investigator, Omer Othman Abdullah, Associate consultant ophthalmologist, Ibinsina Modern Eye and Retina Center
Organization: Ibinsina Modern Eye and Retina Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMER 14
Record Dates: First submitted 2022-02-19; First posted 2022-03-14 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Intraocular Lens Complication
Keywords: Intraocular lens dislocation; Scleral re-fixation; scleral fixation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The scleral pocket for the primary implanted IOL (Other): single arm
  Interventions: Other: The surgical intervention

INTERVENTIONS:
Other: The surgical intervention — The participant's primary IOL is re-fixed without utilizing any new material.

SUMMARY:
To minimize multiple manipulations and to decrease the economical burden; here, we describe how to utilize the patient's own dislocated intraocular lens to re-fixate with the sclera.

DETAILED DESCRIPTION:
When a scleral fixated intraocular lens (IOL) is displaced; routinely it is extracted and exchanged with another IOL and re-fixated to the sclera or another modality can be used. Both can carry many complications due to multiple manipulations. Nevertheless, suture and/or haptic end exposure is another expected future complication, which can range from foreign body sensation to endophthalmitis.

Here, the investigators utilized the same participant's IOL with minimum manipulations and the haptic ends buried inside scleral pockets to prevent future exposure and complications. The pocket entry is sutured with 8/0 vicryl, which is absorbable, to overcome complications.

ELIGIBILITY:
Inclusion Criteria:

* Dislocated primary scleral fixed IOL

Exclusion Criteria:

* Iris claw IOL
* Anterior chamber IOL

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
The slit-lamp examination. | The fourth week post-operatively.
  To assess the intra-ocular pressure mmHg, the re-fixated intraocular lens position ( central, tilted or displaced),and leakage from the incisions, and the hemorrhage ( whether in the anterior segment or in the posterior segment).

SECONDARY OUTCOMES:
The visual acuity. | The fourth week post-operatively.
  To assess both the uncorrected and the best corrected visual acuity ( with glasses).

CONTACTS AND LOCATIONS:
Overall Officials: Omer Abdullah, M.Sc., Principal Investigator — Ibinsina Modern Eye and Retina Center
Locations (1):
- Ibinsina Modern eye and retina center, Erbil, Iraq

IPD SHARING:
Plan to Share IPD: No